CLINICAL TRIAL: NCT06135402
Title: Monocentric, Prospective, Randomised, Single Blinded, Active-controlled Trial to Prove That the Treatment With Monalisa Glide is Equal to Topic Clobetasol Propionate Maintenance Therapy in Vulvar Lichen Sclerosus
Brief Title: Comparison of Laser Treatment With Clobetasol Therapy in Patients With Lichen Sclerosus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Laser-Lichen
Record Dates: First submitted 2023-10-24; First posted 2023-11-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Lichen Sclerosus
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus | interventions — Therapeutics; Clobetasol

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, randomized, single-blinded, active-controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser group (Experimental): 3 monthly fractional laser treatment according to the user manual (correct applicator, vulvar and vaginal preset). In between daily local skin care with a drug free product of patients' choice.
  Interventions: Device: Treatment with Monalisa Glide Laser
- Clobetasol group (Active Comparator): Maintenance treatment with vulvar TCS (clobetasol) application 2x/week. Instruction given at trial start and monthly check up for treatment control Daily local skin care with a drug free product of patients' choice.
  Interventions: Drug: Treatment with Clobetasol

INTERVENTIONS:
Device: Treatment with Monalisa Glide Laser — 3 fractional laser treatment-sessions with Monalisa Glide
  Arms: Laser group
Drug: Treatment with Clobetasol — Application of Clobetasol twice per week
  Arms: Clobetasol group

SUMMARY:
With this trial the investigators look for the effect of Laser maintenance therapy in patients with vulvar lichen sclerosus compared to the maintenance standard treatment clobetasol propionate.

DETAILED DESCRIPTION:
Vulvar Lichen sclerosus (VLS) is a chronic inflammatory cutaneous disorder, which can lead to scarring, impaired sexual function and malignancy. Gold standard treatment is topical corticosteroids (TCS) initially daily for 12 weeks. To avoid new flourishing of the disease a life-long maintenance treatment 2x/week is later recommended. Fractional CO2-Laser has shown a positive effect on vulvovaginal skin quality with improvement of urogenital atrophy and also lichen sclerosus. This randomised trial compares efficacy of laser treatment to TCS maintenance as well as the duration of the laser effect.

ELIGIBILITY:
Inclusion Criteria:

* Pre- or postmenopausal
* 12 weeks of continuous topical clobetasol treatment completed.
* Written informed consent
* German speaking (Study information and IC available only in German)

Exclusion Criteria:

* Contraindication and limitations for the use of Mona Lisa Glide-Laser as described in the instructions for use
* Contraindication for the use of topic clobetasol
* History of vulva laser
* Immune-suppression
* Pregnancy or planned pregnancy, breast feeding.
* Clinically significant concomitant diseases states as severe renal failure, hepatic dysfunction, severe cardiovascular disease, cancer.
* History of vulvar or pelvic radiation therapy
* Uncertain vulvar findings, which require a biopsy.
* Acute vulvitis, especially recurrent genital herpes
* History of vaginal mesh implantation within 6 months preceding this study
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the subject
* Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation
* Previous enrolment into the current investigation
* Enrolment of the PI, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Lichen Score | 3 months
  The difference between the initial Lichen score and the score at 3 month after treatment start = 1 month after EOT

SECONDARY OUTCOMES:
Lichen Score Follow up | 15 months
  Lichen score at 4, 8 and 12 months after EOT, Scale from 0 (no symptoms) to 12 (symptoms)
Vulva assessment Scale | 15 months
  Vulva assessment scale at 1, 4, 8 and 12 months after EOT, Scale from 0 (no symptoms) to 12 (symptoms)
German Pelvic floor questionnaire | 15 months
  Shortened Pelvic floor questionnaire at 1, 4, 8, 12 months after EOT

CONTACTS AND LOCATIONS:
Overall Officials: Gesine Meili, MD, Principal Investigator — Clinic of obstetrics and gynecology
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No